CLINICAL TRIAL: NCT04165798
Title: KEYMAKER-U01 Master Study: A Phase 1/2, Umbrella Study With Rolling Arms of Investigational Agents, Pembrolizumab, and Chemotherapy, Alone or in Combination, in Participants With Non-small Cell Lung Cancer (NSCLC)
Brief Title: KEYMAKER-U01 Umbrella Master Study: Studies of Investigational Agents With Either Pembrolizumab (MK-3475) Alone or With Pembrolizumab PLUS Chemotherapy in Participants With Non-small Cell Lung Cancer (NSCLC) (MK-3475-U01/KEYMAKER-U01)
Status: Recruiting | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3475-U01; MK-3475-U01 (Other: MSD); KEYMAKER-U01 (Other: MSD)
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To identify novel biomarkers, biospecimens (i.e., blood components, tumor material) will be collected to support analyses of cellular components (eg, protein, DNA, RNA, metabolites) and other circulating molecules.
  Investigations may include but are not limited to:
  Tumour tissue analyses, germline (blood) genetic analyses (e.g. single nucleotide polymorphism [SNP] analyses, whole exome sequencing, whole genome sequencing)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective NSCLC Participants: Male and female participants with histologically-confirmed diagnosis of squamous or nonsquamous NSCLC will be screened for participation in 1 of several pembrolizumab substudies.
  Interventions: Diagnostic Test: Tumor Imaging; Procedure: Tumor Tissue Collection; Procedure: Blood Sample Collection

INTERVENTIONS:
Diagnostic Test: Tumor Imaging — Participants will undergo tumor imaging using either a magnetic resonance imaging (MRI) scan or a computed tomography (CT) scan.
Procedure: Tumor Tissue Collection — Participants without archival tumor tissue samples will undergo tumor tissue collection for newly obtained tumor tissue.
Procedure: Blood Sample Collection — Participants will have blood samples drawn for analysis of:
  * genetics
  * ribonucleic acid (RNA)
  * serum biomarker
  * plasma biomarker
  * circulating tumor DNA (ctDNA)

SUMMARY:
This study is referred to as the "umbrella master protocol" for pembrolizumab (MK-3475) in the treatment of non-small cell lung cancer (NSCLC). This pembrolizumab NSCLC umbrella master protocol uses a platform design and consists of this master screening study and additional substudies. Each substudy will enroll a different population of NSCLC participants.

DETAILED DESCRIPTION:
The following pembrolizumab substudies will evaluate the efficacy of different investigational agents in combination with pembrolizumab given in sequence or in combination with pembrolizumab PLUS chemotherapy:

* KEYMAKER-U01 Substudy 01A: A Phase 1/2, Umbrella Study With Rolling Arms of Investigational Agents, With Pembrolizumab With or Without Chemotherapy in Treatment-Naive Participants With Stage IV Non-small Cell Lung Cancer (NSCLC) (MK-3475-01A) - NCT04165070
* KEYMAKER-U01 Substudy 2: A Phase 2, Umbrella Study with Rolling Arms of Investigational Agents in Combination with Pembrolizumab in Treatment Naïve Patients with PD-L1 Positive Advanced Non-small Cell Lung Cancer (NSCLC) (MK-3475-01B) - NCT04165083
* KEYMAKER-U01 Substudy 3: A Phase 2, Umbrella Study with Rolling Arms of Investigational Agents in Combination with Pembrolizumab in Patients with Advanced Non-small Cell Lung Cancer (NSCLC) Previously Treated with anti-PD-(L)1 Therapy (MK-3475-01C) - NCT04165096
* KEYMAKER-U01 Substudy 01E: A Phase 2 Umbrella Study With Rolling Arms of Investigational Agents With or Without Chemotherapy in Combination With Pembrolizumab in Treatment of Participants With Newly Diagnosed Resectable Stages II-IIIB (N2) Non-small Cell Lung Cancer (NSCLC) (MK-3475-01E) - NCT06788912
* KEYMAKER-U01 Substudy 01F: A Phase 1b/2 Umbrella Study With Rolling Arms of Investigational Agents for Second-line Treatment of Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With KRAS G12C Mutations (MK-3475-01F) - NCT number pending
* KEYMAKER-U01 Substudy 01G: A Phase 2, Umbrella Study With Rolling Arms of Investigational Agents in Combination With Pembrolizumab With or Without Platinum-based Chemotherapy in Treatment-Naïve Participants With Stage IV Non-small Cell Lung Cancer (NSCLC) (MK-3475-01G) - NCT06731907
* KEYMAKER-U01 Substudy 01H: A Phase 2, Randomized, Umbrella Study With Rolling Arms of Investigational Agents in Participants with Previously Treated Stage IV Nonsquamous Non-small Cell Lung Cancer (NSCLC) (MK-3475-01H) - NCT06780085
* KEYMAKER-U01 Substudy 01I: A Phase 2, Randomized, Umbrella Study With Rolling Arms of Investigational Agents in Participants With Previously Treated Stage IV Squamous Non-small Cell Lung Cancer (NSCLC) (MK-3475-01I) - NCT06780098
* KEYMAKER-U01 Substudy 01J: A Randomized Phase 2 Umbrella Study With Rolling Arms of Investigational Agents for First-line Treatment of Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With KRAS G12C Mutations (MK-3475-01J) - NCT number pending

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically- or cytologically-confirmed diagnosis of Stage IV squamous or nonsquamous NSCLC
* Has measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants with histologically-confirmed diagnosis of squamous or nonsquamous NSCLC
Sampling Method: Probability Sample
Enrollment: 1065 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2032-02-13 (Estimated); Study Completion 2032-02-13 (Estimated)

PRIMARY OUTCOMES:
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Level: Tumor Proportion Score (TPS) <1% vs. TPS =1% | Up to approximately 1 month
  Participants' tumors will be evaluated for their PD-L1 tumor expression level using archival tumor tissue samples or newly obtained tumor tissue. The percentage of participants who have a Tumor Proportion Score (TPS) <1% vs. a TPS =1% will be presented.
Tumor Histology Status: Squamous Non-small Cell Lung Cancer (NSCLC) vs. Nonsquamous NSCLC | Up to approximately 1 month
  Participants' tumors will be evaluated for their tumor histology status as being either squamous vs. nonsquamous NSCLC using archival or newly obtained tumor tissue samples. The percentage of participants who have squamous vs. nonsquamous NSCLC will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (47):
- United States (18):
  - Banner MD Anderson Cancer Center ( Site 0001), Gilbert, Arizona
  - City of Hope ( Site 0014), Duarte, California
  - UCSF Medical Center at Mission Bay ( Site 0007), San Francisco, California
  - Georgetown University ( Site 0036), Washington D.C., District of Columbia
  - University of Kentucky Markey Cancer Center ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 0003), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0002), Boston, Massachusetts
  - Oncology Hematology West, PC DBA Nebraska Cancer Specialists ( Site 0031), Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center ( Site 0016), Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0037), Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0034), New York, New York
  - Sanford Fargo Medical Center ( Site 0039), Fargo, North Dakota
  - Cleveland Clinic Main ( Site 0006), Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center ( Site 0015), Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania ( Site 0010), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 0038), Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center ( Site 0009), Houston, Texas
- Hungary (3):
  - Petz Aladar Megyei Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 0060), Budapest
- Israel (7):
  - Soroka Medical Center ( Site 0072), Beersheba
  - Rambam Health Care Campus-Oncology ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence, Firenze
  - IRCCS Ospedale San Raffaele ( Site 0171), Milan
  - Policlinico Gemelli di Roma ( Site 0174), Roma
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0152), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Seoul National University Bundang Hospital ( Site 0081), Seongnam-si, Kyonggi-do
  - Severance Hospital ( Site 0080), Seoul
  - Samsung Medical Center ( Site 0082), Seoul
- Spain (3):
  - ICO L Hospitalet ( Site 0090), L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic de Barcelona ( Site 0092), Barcelona
  - Hospital Universitario Quiron Madrid ( Site 0091), Madrid
- Taiwan (3):
  - Changhua Christian Hospital ( Site 0181), Changhua
  - Taipei Medical University Hospital ( Site 0180), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0182), Taoyuan District
- Ukraine (4):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 0463), Cherkasy, Cherkasy Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical Oncological Center" of Ivano-Frankivsk Reg ( Site 0460), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 0461), Rivne, Rivne Oblast
  - Uzhhorod Multispecialty City Clinical Hospital ( Site 0462), Uzhhorod, Zakarpattia Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/